CLINICAL TRIAL: NCT04914169
Title: The Intelligent Cardiopulmonary Rehabilitation System: A Feasibility Study in Healthy Subjects
Brief Title: The Intelligent Cardiopulmonary Rehabilitation System: A Feasibility Study
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Yen-Nung Lin, Director of Physical Medicine and Rehabilitation, Taipei Medical University WanFang Hospital
Other Study IDs: N202010010
Record Dates: First submitted 2021-05-24; First posted 2021-06-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Cardiac Rehabilitation
Keywords: cardiac rehabilitation; cardiorespiratory fitness; aerobic exercise; endurance training

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Indoor cycling training: 8 subjects were asked to complete indoor cycling training, 3 times a week for 4 weeks. Each session of training consisted of 30-minute stationary biking (5 minutes of warm-up, 20 minutes of training and 5 minutes of cooldown).
  Interventions: Device: ICRS

INTERVENTIONS:
Device: ICRS — The ICRS enables a stationary bike to automatically adjust the pedaling resistance (i.e. training intensity) according to the subject's heart rate. The training intensity is determined by monitoring whether the subject is able to maintain a 50-70 cycles/min cadence with 60-80% HRR. Subjects heart rate was detected by a wearable device for heart rate, synching with the stationary bike.

SUMMARY:
The Intelligent Cardiopulmonary Rehabilitation System (ICRS) was developed to automatically control the resistance of pedaling in combination with the conventional stationary bike by monitoring the user's heart rate for clinical use. To test its feasibility, 8 healthy participants were recruited to complete 12 sessions (3 times per week for 4 weeks) of indoor cycling on the stationary bicycle with ICRS. Subjects were received cardiopulmonary exercise testing (CPET) before and after the biking sessions.The 60-80% of heart rate reserve (HRR) of each participant was determined according to their first CPET results. The algorithm of ICRS was designed to enable the bicycle to adjust its training intensity in accordance with the subject's 60-80% HRR which was detected by wearing a wristband heart rate monitor during cycling. With ICRS, the participants' heart rates during training were expected to fall in the 60-80% HRR, increasing their cardiopulmonary fitness after 12 sessions of indoor cycling.

ELIGIBILITY:
Inclusion Criteria:

* age of 20-50
* no regular exercise habits
* no documented cardiopulmonary disease

Exclusion Criteria:

* abnormal lung function
* medications affecting exercise capacity
* hypertension
* diabetes mellitus
* recent illness including upper respiratory tract infection
* the presence of any factor that may limit ability to participate in the CPET

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy subjects
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Peak oxygen consumption (VO2-peak) | 4 weeks
  Oxygen consumption (VO2- peak) were measured during our cardiopulmonary test (with a incremental biking and a gas analyzer). The workload was increased at a ramp rate of 5-10 W/min. A cadence at 50~70 rpm was to be maintained.

SECONDARY OUTCOMES:
Peak workload | 4 weeks
  The peak workload is measured during a the cardiopulmonary exercise test with a ramped stationary biking.
Compliance of training during the training sessions | 4 weeks
  The percentage of time that a subject's heart rate falls in his or her estimated 60-80% HRR over the 12 sessions of training.
Averaged workload during the training sessions | 4 weeks
  The averaged workload (watt) that a subject paddled on the stationary bike over the 12 sessions of training.

CONTACTS AND LOCATIONS:
Locations (1):
- Wan Fan Hospital, Taipei, Taiwan